CLINICAL TRIAL: NCT05983783
Title: A Prospective Randomized Controlled Study Comparing the Efficacy and Safety of Rezvilutamide+ADT+Docetaxel Versus Rezvilutamide +ADT in the Treatment of Patients With Metastatic Hormone-sensitive Prostate Cancer (mHSPC)
Brief Title: Comparing the Efficacy and Safety of Rezvilutamide+ADT+Docetaxel Versus Rezvilutamide +ADT in the mHSPC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hua Lixin, M.D., The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-SR-376
Record Dates: First submitted 2023-08-02; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Metastatic Prostate Cancer; Hormone Sensitive Prostate Cancer; Chemotherapy Effect
Keywords: Rezvilutamide; mHPSC; chemotherapy; Androgen deprivation therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rezvilutamide+ADT+Docetaxel (Experimental): Rezvilutamide: 240 mg (3 tablets of 80 mg each) orally once daily (QD), can be taken with or without food.
  Docetaxel 6 cycles
  Interventions: Drug: Docetaxel
- Rezvilutamide+ADT (Active Comparator): Rezvilutamide: 240 mg (3 tablets of 80 mg each) orally once daily (QD), can be taken with or without food.
  Interventions: Drug: Rezvilutamide

INTERVENTIONS:
Drug: Docetaxel — This is Triple drug regimen for mHSPC
  Other Names: Rezvilutamide
  Arms: Rezvilutamide+ADT+Docetaxel
Drug: Rezvilutamide — This is doubling drug regimen for mHSPC
  Other Names: ADT
  Arms: Rezvilutamide+ADT

SUMMARY:
Evaluate whether the combination of Rezvilutamide and androgen deprivation therapy (ADT) with docetaxel improves overall survival (OS) in patients with metastatic hormone-sensitive prostate cancer (mHSPC) compared to the combination of Rezvilutamide and ADT.

DETAILED DESCRIPTION:
To investigate the value of chemotherapy in the treatment of high-burden of mHSPC on the background of next-genertion of AR inhibitors.

ELIGIBILITY:
Inclusion Criteria:

1. Males aged ≥40 years and ≤80 years.
2. Histologically or cytologically confirmed prostate adenocarcinoma.
3. Metastatic disease.
4. Eligible for ADT and Docetaxel.
5. Started or not started first-generation androgen deprivation therapy (ADT), but not exceeding 12 weeks before randomization.
6. ECOG score of 0 or 1.
7. Laboratory tests meet the following requirements:

   * Hematology: neutrophils ≥1.5×10^9/L, platelets ≥100×10^9/L, hemoglobin ≥9g/dL.
   * Renal function: serum creatinine ≤1.5× upper limit of normal (ULN).
   * Liver function: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5× ULN, total bilirubin (TBIL) ≤1.5× ULN.
   * Coagulation function: international normalized ratio (INR) <1.5.
8. Study subjects: Patients with mHSPC have a confirmed pathology of prostate adenocarcinoma with high tumor burden, which is defined by having at least one of the following conditions:

1) Bone scan showing ≥4 bone metastatic lesions (with at least one site outside the pelvis or spine).

2) CT/MRI revealing visceral metastatic lesions (excluding lymph nodes).

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible to participate in this study:

1. Prior use of LHRH agonists/antagonists; second-generation androgen receptor (AR) inhibitors such as enzalutamide, ARN-509, darolutamide (ODM-201), or other investigational AR inhibitors; CYP17 enzyme inhibitors such as abiraterone acetate or oral ketoconazole for anti-tumor treatment of prostate cancer; chemotherapy or immunotherapy for prostate cancer prior to randomization.
2. Received radiation therapy/radiopharmaceutical treatment within 2 weeks before randomization.
3. Any of the following conditions within 6 months before randomization: stroke, myocardial infarction, severe/unstable angina pectoris, coronary artery/peripheral artery bypass surgery, congestive heart failure (New York Heart Association class III or IV).
4. Previous malignancy, except adequately treated basal cell carcinoma or squamous cell carcinoma of the skin or superficial bladder cancer not invading the deeper muscle layer (i.e., pTis, pTa, and pT1) and any other cancer in complete remission for at least 5 years before randomization.
5. Gastrointestinal diseases or procedures that are expected to significantly interfere with the absorption of study treatment.
6. Inability to take oral medication.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
rPFS | 36 months
  radiographic Progression-Free Survival

SECONDARY OUTCOMES:
prostate-specific antigen (PSA) response rate | 36 months
  percentage of patients with a decreasing PSA following the regimens discussed above
time to castration-resistant prostate cancer (CRPC) | 36 months
  time to PSA progression

OTHER OUTCOMES:
time to next bone-related event | 36 months
  Including bone structure, pain, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Lixxin Hua, Principal Investigator — Urology Dpt, First Affiliated Hospital of Nanjing Medical University
Locations (1):
- Urology dpt, First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-08-02): https://cdn.clinicaltrials.gov/large-docs/83/NCT05983783/Prot_ICF_000.pdf